CLINICAL TRIAL: NCT06900946
Title: Evaluation of the Effects of Gluten Free Diet on Clinical Symptoms and Glycemic Index in Type 2 Diabetic Patients With Non-celiac Gluten Sensitivity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Prof., National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 43012148
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Non Celiac Gluten Sensitivity
Keywords: Type 2 Diabetes; T2DM; NCGS; Non celiac gluten sensitivity; Gluten free diet; GFD
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glutens; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): 3 grams of gluten powder taken daily
  Interventions: Other: gluten
- Control (Placebo Comparator): 3 grams of corn starch powder taken daily
  Interventions: Other: cornstarch

INTERVENTIONS:
Other: gluten — The intervention group will receive 3 grams of gluten powder daily
  Arms: Intervention
Other: cornstarch — The control group will receive 3 grams of cornstarch powder daily
  Arms: Control

SUMMARY:
Confirmed cases of type 2 diabetes who have presented with gastrointestinal symptoms and have no diagnosed gastrointestinal diseases will be referred to the laboratory for testing of tTG IgA and total IgA antibodies to rule out celiac disease, as well as IgE antibody testing to exclude wheat allergy. After ruling out celiac disease, wheat allergy, and irritable bowel syndrome (IBS) using the Rome IV criteria, the patients will be invited to the clinic. The study's objectives, methods, and procedures will be explained, and written informed consent will be obtained from patients who are willing to participate.

At the start of the study, each patient's weight will be measured while wearing light clothing using a mechanical scale (with an accuracy of 100 grams), and height will be measured without shoes using a wall-mounted meter (with an accuracy of 0.5 cm). The body mass index (BMI) of the patients will then be calculated. Additionally, general patient information will be recorded on the data collection form, and the gastrointestinal symptoms questionnaire (NCGS-SQ) will be completed.

Next, blood sample will be drawn from the patients after fasting for 8 to 12 hours, and their serum will be collected to measure glycemic indices, including FBS, HbA1c, insulin, and HOMA-IR. A gluten-free diet (GFD) will be designed by a nutritionist to maintain the weight of type 2 diabetic patients and must be followed for 6 weeks. Carbohydrate distribution and diabetes-related recommendations will also be provided for the patients.

Patient follow-up will be conducted via phone calls to ensure adherence to the diet and to prevent sample loss. Diet compliance will be assessed by a nutritionist, who will review the intake of any gluten-containing foods.

After six weeks (Phase 1), glycemic indices will be re-evaluated through blood tests. Patients who have adhered to the diet optimally and experienced significant improvement in gastrointestinal symptoms will be suspected of having NCGS. If they agree, they will remain in the study and participate in a double-blind, placebo-controlled randomized trial. Those who do not show improvement in gastrointestinal symptoms during the first six weeks will be excluded from the study.

In Phase 2, both the patients and the researchers assessing them will be blinded to the treatment being studied. Intervention group (gluten group) will receive 3 grams of gluten, and control group (placebo group) will receive 3 grams of corn starch powder, to be consumed daily mixed with milk or another beverage. Patients in both groups will continue following their gluten-free diets. At the end of study , glycemic indices will be re-evaluated, and changes in those indices over the 6-week period will be assessed. Additionally, a clinical symptoms questionnaire will be completed via phone calls every three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Exclusion of Celiac Disease and Wheat Allergy (tTG IgA antibody test for celiac disease exclusion and IgE antibody test for ruling out wheat allergy)
* Exclusion of Irritable Bowel Syndrome (IBS) using the Rome IV diagnostic criteria by a gastroenterologist
* No adherence to any specific diet in the past 6 months, including the gluten-free diet (GFD)
* Willing and capable of following a gluten-free diet (GFD)
* No consumption of alcohol or drugs
* No use of corticosteroids or antidepressant medications
* No history of thyroid disorders, autoimmune diseases, cancer, or gastrointestinal diseases

Exclusion Criteria:

* Inability or unwillingness to continue with the study
* Pregnancy or Lactation
* Occurrence of any side effects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | Initially, week 6, and week 12
  HbA1C change from baseline
Fasting Blood Sugar (FBS) | Initially, week 6, and week 12
  Blood sugar change from baseline
Insulin | Initially, week 6, and week 12
  blood insulin change from baseline
Clinical symptoms | Initially, week 3, week 6, week 9, and week 12
  changes in GI clinical symptoms from baseline according to visual analogue score of 0-10

SECONDARY OUTCOMES:
HOMA-IR | Initially, Week 6, and Week 12
  HOMA-IR change from the baseline
Abdominal pain or discomfort | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in abdominal pain from baseline according to visual analogue score of 0-10
Heartburn | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in heart burn symptom from baseline according to visual analogue score of 0-10
Acid reflux | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in sense of acid reflux from baseline according to visual analogue score of 0-10
Nausea and vomiting | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in nausea and vomiting symptoms from baseline according to visual analogue score of 0-10
Bloating | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in bloating sense from baseline according to visual analogue score of 0-10
Borborygmus (stomach rumbling) | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in Borborygmus symptoms from baseline according to visual analogue score of 0-10
Abdominal distension | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in abdominal distension symptoms from baseline according to visual analogue score of 0-10
Feeling of belching (burping) | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in feeling of belching from baseline according to visual analogue score of 0-10
flatulence | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in flatulence symptom from baseline according to visual analogue score of 0-10
Reduced stool passage | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in feeling reduced stool passage from baseline according to visual analogue score of 0-10
Increased stool passage | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in feeling increased stool passage from baseline according to visual analogue score of 0-10
Loose stools | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in number of loose stools per day from baseline according to visual analogue score of 0-10
Hard stools | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in hard stools per day from baseline according to visual analogue score of 0-10
Urgency to defecate | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in frequency of urgency to defecate from baseline according to visual analogue score of 0-10
Feeling of incomplete evacuation | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in feeling of incomplete evacuation from baseline according to visual analogue score of 0-10
Extraintestinal symptoms | Initially, Week 3, Week 6, Week 9, and Week 12
  changes in extra-intestinal symptoms from baseline according to visual analogue score of 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Behboud Clinic, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided